CLINICAL TRIAL: NCT04441385
Title: Bicentric, Phase 2, Randomized, Open-label Study to Evaluate the Efficacy and Safety of Maraviroc Associated With Standard Treatment in Hospitalized Patients With Pulmonary SARS-CoV-2 Infection (COVID-19).
Brief Title: Study to Evaluate the Efficacy and Safety of Maraviroc in SARS-CoV-2 Infection (COVID-19).
Acronym: MARACOVID
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: lack of viability
Sponsor: Hospital Universitario Infanta Leonor (Other)
Collaborators: Hospital Clinic of Barcelona (Other); ViiV Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MARACOVID; 2020-002011-21 (EudraCT Number)
Record Dates: First submitted 2020-06-18; First posted 2020-06-22 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2020-07

CONDITIONS: COVID-19
Keywords: SARS-CoV-2; ARDS; Acute respiratory distress syndrome; maraviroc
MeSH Terms: conditions — COVID-19; Respiratory Distress Syndrome | interventions — Maraviroc

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Test arm (Experimental): 100 subjects will be randomly assigned to this arm. Patients in the test group will receive 300 mg of maraviroc BID for 14 days (added to standard care).
  Interventions: Drug: Maraviroc 300 mg
- Control arm (Other): 100 subjects will be randomized in this arm and will be treated according to the standard care. The Ministry of Health has issued detailed guidelines for the management of COVID-19. Local Institutional Guidelines and Protocols for supportive management will also be implemented.
  Interventions: Other: Standard care therapy

INTERVENTIONS:
Drug: Maraviroc 300 mg — Patients will receive maraviroc 300 mg twice daily for 14 days
  Other Names: Celsentri; Selzentry
  Arms: Test arm
Other: Standard care therapy — Subjects randomized to control group will be on standard care treatment according to the Ministry of Health and Local Guidelines and Protocols.
  Arms: Control arm

SUMMARY:
This is a bicentric, phase 2, randomized, open-label study to evaluate the efficacy and safety of maraviroc associated with standard treatment in hospitalized patients with pulmonary SARS-CoV-2 infection (COVID-19).

DETAILED DESCRIPTION:
This is a bicentric, phase 2, randomized, open-label study to evaluate the efficacy and safety of maraviroc associated with standard treatment in hospitalized patients with pulmonary SARS-CoV-2 infection (COVID-19), to prevent disease progression to severe Acute Respiratory Distress Syndrome (ARDS).

Patients will be randomized to receive maraviroc (300 mg BID for 14 days) plus standard treatment, or standard treatment alone.

200 subjects will be enrolled and randomized 1:1 in this study.

ELIGIBILITY:
Inclusion Criteria:

* 1. Male or female adult ≥ 18 years of age at the time of giving informed consent.
* 2. Subject is hospitalized.
* 3. SARS-CoV-2 infection confirmed by PCR or other commercial or public health tests, in any biological sample obtained up to 4 days prior to randomization, or that meets locally accepted criteria for clinical diagnosis of COVID-19.
* 4. Lung involvement confirmed by at least one of the following criteria:

  1. Radiological infiltrates on imaging test (conventional radiography, computed tomography (CT) or other)
  2. In the absence of radiological infiltrates, an SpO2 < 95% without oxygen supporting therapy (breathing ambient air), combined with cough, crackles on physical exam, or an LDH > 300 U/L with no other cause.
* 5. Symptom onset ≤ 8 days prior to randomization.
* 6. Understands and agrees to comply with planned study procedures.
* 7. Women of childbearing potential must have a negative test for pregnancy (blood or urine) before their inclusion and agree to use an accepted method of contraception for the duration of the study.
* 8. Subject (or legally authorized representative) provides written informed consent prior to initiation of any study procedures.

Exclusion Criteria:

* 1. SpO2 ≤ 91% breathing ambient air and SpO2 < 95% with oxygen in nasal cannula at 2 lpm.
* 2. Patient's attending physician considers the study is not the best medical option, or follow-up after discharge will be difficult.
* 3. A patient who, in the investigator's opinion, is unlikely to survive > 48 hours from inclusion in the study.
* 4. Patients with severe chronic kidney disease (ClCr < 30 ml/min/1.73 m2 or receiving renal replacement therapy in any of its modalities).
* 5. Severe liver disease (Child-Pugh C, ALT > 5 times above upper limit of normal (LSN).
* 6. COPD with FEV1 < 70.
* 7. Known active neoplasia.
* 8. HIV infection. Patients with known HIV infection, under follow-up, and immunovirological stability (CD4> 500 and undetectable viral load) for at least 6 months before inclusion in this study may be included.
* 9. Hemoglobin < 9 gr/dL.
* 10. Prolonged QT, defined as a QT interval > 460 ms. (or > 450 ms. in case of family history of sudden death or long QT syndrome or personal history of repeat syncope without an etiological diagnosis). This criterion will only apply if the standard treatment contains drugs with an effect on the duration (prolongation) of the QT interval.
* 11.Significant cardiovascular disease, including:

  1. History of acute myocardial infarction, acute coronary syndrome (unstable angina, coronary by-pass surgery, angioplasty, or coronary stenting) ≤ 6 months prior to randomization
  2. Symptomatic heart failure (NYHA grade 2 or more) history, or current evidence of cardiac arrhythmia (except atrial fibrillation or flutter and paroxysmal supraventricular tachycardia) and/or conduction abnormalities (excluding branch blocks or Wenckebach grade I and II atrioventricular blocks).
* 12. Known or suspected active autoimmune disease
* 13. Pregnancy or breastfeeding, or positive pregnancy test at baseline or screening visit
* 14. Patients who are expected to be transferred to another facility sooner than 72 hours after inclusion in the study.
* 15. Patients who have received experimental treatment (off-label, compassionate use, or in clinical trials) within 30 days prior to the screening visit, except for treatment considered standard initiated on admission to hospital, up to 48 hours before inclusion in the study.
* 16. Patients who have a history of allergic reactions to maraviroc or any of its components.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-06-26 (Actual); Primary Completion 2021-02-08 (Actual); Study Completion 2021-02-08 (Actual)

PRIMARY OUTCOMES:
Proportion of patients developing severe ARDS. | 28 days
  A patient with a saturation of 90% or less despite the use of a reservoir mask without rebreathing with a flow of 7 liters per minute (FiO2 0.6 or higher), will be considered to have severe ARDS. These oximetric criteria have a close correlation with a PaO2 / FiO2 of 100 or less, which defines severe ARDS.

SECONDARY OUTCOMES:
All-cause mortality. | 28 days
Percentage of patients requiring tracheal intubation, use of Non-invasive Ventilation NIV or High Flow Nasal Cannula (HFNC) devices during the study period | 28 days
Percentage of patients who progress to severe ARDS, death or ICU admission. | 28 days
Differences in Time to Clinical Improvement | 28 days
  Defined as the time (in hours) from the start of the treatment under study to the normalization of temperature, normalization of respiratory rate and SpO2.
  1. Axillary temperature < 37.5ºC (oral < 37.2ºC) for 48 hours, without antipyretic treatment.
  2. Breathing rate < 24 rpm during the clinical evaluation and at least two consecutive daily evaluations (48 hours).
  3. SpO2 > 93% breathing ambient air during clinical assessment and at least two consecutive daily assessments (48 hours).
Change in clinical status of subject on a 7-point ordinal scale. | 28 days
  The ordinal scale of 7 categories of patient health status ranges from:
  1. Death.
  2. Hospitalized, with invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO).
  3. Hospitalized, with non-invasive ventilation or high flow oxygen devices.
  4. Hospitalized, requiring supplemental oxygen.
  5. Hospitalized, not requiring supplemental oxygen.
  6. Non-hospitalized, activity limitation.
  7. Non-hospitalized, no activity limitation.
Percentage of patients requiring immunosuppressive/immunomodulatory treatment as a rescue medication. | 28 days
Proportion of patients developing adverse effects, serious adverse reactions, laboratory or physical examination findings, EKG abnormalities acquired during the trial, death and adverse events leading to early discontinuation of treatment. | 28 days
  Classification according to the WHO toxicity scale

CONTACTS AND LOCATIONS:
Overall Officials: Víctor Domínguez, MD, Principal Investigator — Hospital Universitario Infanta Leonor
Locations (2):
- Spain (2):
  - Hospital Clínic, Barcelona
  - Hospital Universitario Infanta Leonor, Madrid